CLINICAL TRIAL: NCT01289951
Title: Phase I, Open Label, Unicentric Study of Multiple-dose Pharmacokinetics of Raltegravir in Patients Infected With Human Immunodeficiency Virus and Hepatitis C Virus With and Without Advanced (Child-Pugh C) Hepatic Cirrhosis.
Brief Title: Pharmacokinetic Study of Raltegravir in Human Immunodeficiency Virus/Hepatitis C Virus (HIV/VHC) Coinfected Patients With Advanced (Child-Pugh C) Hepatic Cirrhosis
Acronym: LIVERAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIVERAL
Record Dates: First submitted 2011-02-01; First posted 2011-02-04 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Human Immunodeficiency Virus; Hepatitis C
Keywords: HIV; VHC; Advanced hepatic cirrhosis; Pharmacokinetic; Raltegravir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with Child-Pugh C hepatic-cirrhosis. (Experimental): VIH/VHC coinfected patients with advanced (Child-Pugh C) hepatic cirrhosis.
  Interventions: Drug: Raltegravir 400 mg/12hours
- VIH/VHC coinfected patients without liver damage. (Active Comparator)
  Interventions: Drug: Raltegravir 400 mg/12hours

INTERVENTIONS:
Drug: Raltegravir 400 mg/12hours
  Arms: VIH/VHC coinfected patients without liver damage.
Drug: Raltegravir 400 mg/12hours
  Arms: Patients with Child-Pugh C hepatic-cirrhosis.

SUMMARY:
Raltegravir is the first integrase inhibitor used in humans. It has been shown to be highly efficacious and well tolerated in phase III clinical trials in multidrug experienced human immunodeficiency virus(HIV)-infected patients, as well as initial therapy in untreated patients. Pharmacokinetic studies in healthy adult subjects indicate that the major mechanism of clearance of the drug is glucuronidation mediated by UGT1A1, with a minor contribution of renal excretion of unchanged parent compound. Unlike CYP-based metabolism, glucuronidation is generally found to be relatively unaffected by hepatic disease. A single dose pharmacokinetic study of raltegravir in patients with mild to moderate hepatic insufficiency (Steigbigel et al. 2008) found no clinically important effect on the drug pharmacokinetic profile, with no dosage adjustment being necessary. The liver safety and tolerability of boosted atazanavir (ATV/r) has been evaluated in human immunodeficiency virus and hepatitis C virus (HIV/HCV) coinfected patients with advanced liver disease (decompensated cirrhosis) (Hermida JM et al. 4th IAS: Sidney, 2007). Similar to Raltegravir, ATV is also mainly metabolized by conjugation through UGT1A1. There is an urgent need for potent and efficacious ARV drugs with a clean safety liver profile even in patients with severe liver disease. The investigators hypothesized that pharmacokinetics will not be altered in HIV/HCV patients with advanced (Child-Pugh grade C) cirrhosis or in those with no histologic liver damage.

ELIGIBILITY:
Inclusion Criteria:

* Adults, clinically stable HIV/HCV coinfected patients on HAART with controlled viremia (<50 copies/ml) for at least 6 months. HAART will be based on a boosted protease inhibitor (lopinavir, fosamprenavir or darunavir). Hepatic Stability is defined by the absence of new events of descompensation (Child-Pugh score) in the previous six weeks with no data of progressive hepatic insufficiency.
* Liver biopsy performed during the previous year showing no liver damage (F0-F1 in the Metavir score) or by elastometry results ≤ 6 Kpa, to classify patients in group B.
* Liver cirrhosis guided by biopsy (F4 in the Metavir score) or elastometry: results ≥ 14 Kpa, to classify patients in group A.
* Body mass index (BMI) in the range of 19-35 kg/m2.

Exclusion Criteria:

* HBV surface antigen positive.
* Clinical demonstration of a new descompensation event in the previous 6 weeks.
* Alcohol abuse as an average daily consumption > 20g.
* Treatment with boosted atazanavir, saquinavir or indinavir.
* Concomitant treatment with phenytoin, phenobarbital and rifampinor other UGT1A1 inhibitors.
* Use of any investigational agents (other than ART on expanded access) within 90 days of randomization.
* Active or previous HCV treatment with Ribavirin and /or Peg-interferon if sustained virological response achieved.
* Women taking oral contraceptives
* Pregnancy and lactancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The area under the curve (AUC0-12) calculated from plasma concentrations, the maximum concentration (Cmax) and the the minimum concentration (Cmin) of Raltegravir 400 mg/12 hours in the steady state for both arms. | On the fifth day of treatment with raltegravir
  On the fifth day of treatment, patient will be hospitalized in the clinical trial unit in order to obtaine plasma concentrations previous to the administration of the corresponding dose (basal) and at the following times post-administration: 30min, 1h, 1h30min, 2h, 3h, 4h, 6h, 8h, and 12h. With these measures, (AUC0-12), Cmax and Cmin will be calculated in order to describe the pharmacokinetic of Raltegravir 400 mgBID in the steady state in both arms

SECONDARY OUTCOMES:
Change from baseline in hematology and biochemistry parameters at day 5 and 15, number of adverse events (serious and non serious) notified and number of patients who discontinue the study (drop-out rate). | On day 1, 5 and 15
  Hematology and biochemistry parameters, adverse events notified during the study and drop-out rate will be recorded in order to evaluate the safety and tolerability of multiple doses of raltegravir in HIV/HCV coinfected patients, with no liver damage and with advanced cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Moreno Guillen, MD, Principal Investigator — Hospital Universitario Ramón y Cajal. Madrid
Locations (1):
- Hospital Universitario Ramón y Cajal., Madrid, Madrid, Spain

REFERENCES:
- [Derived] Hernandez-Novoa B, Moreno A, Perez-Elias MJ, Quereda C, Dronda F, Casado JL, Madrid-Elena N, Aguilar M, Fumero E, Molto J, Moreno S. Raltegravir pharmacokinetics in HIV/HCV-coinfected patients with advanced liver cirrhosis (Child-Pugh C). J Antimicrob Chemother. 2014 Feb;69(2):471-5. doi: 10.1093/jac/dkt386. Epub 2013 Oct 4. PMID 24097843